CLINICAL TRIAL: NCT04541446
Title: Study Dynamic Haptic Robotic Trainer (DHRT) and DHRT+ for CVC Insertion Training for Surgical Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Scarlett Miller, Professor, Engineering, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00012206; R01HL127316 (NIH)
Record Dates: First submitted 2020-08-24; First posted 2020-09-09 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Central Line Complication; Central Line Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Residents to receive Dynamic Haptic Robotic Training (Experimental)
  Interventions: Other: Dynamic Haptic Robotic Trainer (DHRT)
- Residents to receive Advanced Dynamic Haptic Robotic Training (Experimental)
  Interventions: Other: Advanced Dynamic Haptic Robotic Trainer (DHRT+)

INTERVENTIONS:
Other: Dynamic Haptic Robotic Trainer (DHRT) — Device trains medical residents to safely perform the needle insertion portion of Central Venous Catheterization.
  Arms: Residents to receive Dynamic Haptic Robotic Training
Other: Advanced Dynamic Haptic Robotic Trainer (DHRT+) — Device offers whole procedural training for medical residents to safely perform the procedure of Central Venous Catheterization.
  Arms: Residents to receive Advanced Dynamic Haptic Robotic Training

SUMMARY:
Human participants will include medical residents. Each year the entering 1st year medical residents at Hershey Medical Center and Cedars-Sinai Medical Center will be taught to perform these procedures using the DHRT or the DHRT+ devices. The resident's performance will be measured and evaluated by these devices during the training. The technique of the training does not differ from what is currently taught at either of these institutions. In addition the residents will be required to pass the same skills assessment currently required at their institution. Upon successfully passing the skills assessment the residents will perform CVC interventions on under supervision. After the procedure the investigators will examine patient files to determine any changes in central line related complications and infection rates due to new clinical educational practices.

ELIGIBILITY:
Inclusion Criteria:

* new resident undergoing central venous catheterization training

Exclusion criteria:

* not a new resident undergoing central venous catheterization training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Central Line Related Complications due to new Resident Central Line Training Procedures | baseline (pre-intervention), post-intervention
  Through patient files complication rates will be measured through study completion, an average of one year after having procedure performed.
Change in Central Line Related Infections due to new Resident Central Line Training Procedures | baseline (pre-intervention), post-intervention
  Through patient files post procedural infection rate is measured through study completion, an average of one year after having procedure performed.

CONTACTS AND LOCATIONS:
Overall Officials: Scarlett R Miller, Ph.D., Principal Investigator — Penn State University; Jason Z. Moore, Ph.D., Principal Investigator — Penn State University
Locations (2):
- United States (2):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Hershey Medical Center, Hershey, Pennsylvania